CLINICAL TRIAL: NCT06983639
Title: FIT Versus Colonoscopy for Post-polypectomy Surveillance
Brief Title: Randomized Trial Comparing Fecal Testing (FIT) to Colonoscopy for Post-polypectomy Surveillance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Sykehuset Ostfold (Other); University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); Sykehuset Telemark Hospital Trust (Unknown); Helse Møre og Romsdal HF (Other Government); St. Olavs Hospital (Other); University Hospital of Northern Norway, Tromsø, Norway (Unknown); Sykehuset i Vestfold HF (Other); Helse Stavanger HF (Other Government); Turku University Hospital (Other Government); Helsinki University Central Hospital (Other); Randers Regional Hospital (Other); Viborg Regional Hospital (Other); Gødstrup Hospital (Other); Horsens Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 744836
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms
Keywords: surveillance; polyp
MeSH Terms: conditions — Colorectal Neoplasms; Polyps | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopy (Active Comparator): Colonoscopy surveillance after polyp removal
  Interventions: Diagnostic Test: Colonoscopy
- Fecal blood testing (Experimental): Fecal testing as surveillance after polypectomy
  Interventions: Diagnostic Test: Fecal occult blood testing

INTERVENTIONS:
Diagnostic Test: Fecal occult blood testing — Fecal testing for blood as surveillance efter polyp removal
  Arms: Fecal blood testing
Diagnostic Test: Colonoscopy — Colonoscopy after polyp removal according to guidelines
  Arms: Colonoscopy

SUMMARY:
From observational studies, it is know that the risk of developing colorectal cancer after polyp removal is lower if the patients adheres to surveillance recommendations. However, colonoscopy is burdensome for patients and colonoscopy availability is limited in many parts of the world. In addition, more than half of surveillance colonoscopies are without any findings. The trial investigates whether surveillance using fecal testing for blod is as good as colonoscopy after removal of colorectal polyps.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in the world and develops from benign colorectal polyps. Colonoscopy with polyp removal reduces colorectal cancer incidence and mortality. Patients who have had polyps removed are at increased risk for metachronous polyps and subsequent cancer and are referred to colonoscopic surveillance at regular intervals, the first one usually scheduled three years after polypectomy. Today, these comprise 15-25% of all colonoscopies, but in >85%, no high-risk pathology is found. Thus, post-polypectomy surveillance consumes major resources without benefit to the patients, and these resources are much needed for colonoscopies due to other indications in an aging population. Additionally, colonoscopy requires burdensome bowel-cleansing, discomfort during the examination, absenteeism from work and sometimes need for an escort. Severe complications like bleeding and perforation may occur. Overdiagnosis and overtreatment of benign lesions occur in a large proportion of examinations as most polyps will never develop into colorectal cancer, even if left untreated.

Sensitive fecal occult blood tests (FIT) have been developed that may detect colorectal cancer with the same sensitivity as colonoscopy. The test is cheap, is easily distributed by mail and may be performed at home. If the test detects blood, colonoscopy is indicated. FIT has been used in colorectal screening program for years, but has not yet been thoroughly investigated for post-polypectomy surveillance purposes.

The trial is a pragmatic non-inferiority randomized trial in which patients who are eligible for 3-year colonoscopic surveillance are offered either colonoscopy (standard care) or FIT followed by a colonoscopy in case of a positive test result (Figure 1). FIT may decrease colonoscopy surveillance demand by > 50%, which equals a cost saving of almost 30,000,000 Norwegian kroner annually. By proposing FIT for post-polypectomy surveillance, the trial introduce decentralized and personalized medical follow-up of these patients, and at the same time reduce work-absenteeism, patient discomfort, risk of complications and importantly: overdiagnosis and overtreatment of benign colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* High-quality baseline colonoscopy with adequat cleansing and cecal intubation
* Remocval of at least one advanced adenoma
* Clean colon (all polyps removed)
* Signed informed consent

Exclusion Criteria:

* Colorectal cancer
* History of surgical colon resection for any reason
* Genetic cancer syndrome (adenomatous or serrated polyposis syndrome; Lynch or Lynch-like syndrome)
* ≥ 10 adenomas at baseline colonoscopy (cumulative)
* History of advanced serrated lesion, defined as SSL≥ 10mm or with dysplasia
* Inflammatory bowel disease
* On-going palliative care for any reason

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer incidence | 12 years from randomization

SECONDARY OUTCOMES:
Colorctal cancer mortality | 12 years from randomization
Advanced neoplasia incidence | 3 years from randomization
  Findings of colorectal cancer and high-risk polyps
Findings at colonoscopy | 12 years from randomization
  Pathology detected during colonoscopy in both arms
Colonoscopy utilization | 12 years after randomization
  Number of colonoscopies performed
Adherence | 12 years from randomization
  Adherence with colonoscopy and FIT surveillance recommendations. Proportion of participants in each arm who are invited for colonoscopy or FIT surveillance and who actually adheres submit the FIT/undergo colonoscopy.
Cost-effectiveness | 12 years from randomization
  Total cost for FIT-surveillance and colonoscopy surveillance will be calculated and compared, including reimbursement (FIT, colonoscopy, pathology assessment), payment from patients, travel, absenteism from work, cost of complications etc.
Adverse events | 30 days after colonoscopy
  Adverse events after colonoscopy
Carbon footprint | 12 years after randomization
  The carbon footprint in each arm will be calculated and compared. Carbon footprint is the total carbon emission from manufacturing, shipping, use, prosessing, litter-handling etc
FIT accuracy | 3 years after randomization
  Sensitivity, specificity, postive predictive value and negative predicitive value for colorectal cancer and advanced neoplasia at different FIT-thresholds

CONTACTS AND LOCATIONS:
Locations (1):
- Sørlandet sykehus HF, Arendal, Agder, Norway

IPD SHARING:
Plan to Share IPD: No